CLINICAL TRIAL: NCT02044809
Title: A Phase IIa/b, Randomised, Double-blind, Placebo-controlled, Single-site, Parallel Group Clinical Trial to Examine Cannabidiol (CBD) as a Pharmacological Treatment for Cannabis Dependence.
Brief Title: Cannabidiol: a Novel Intervention for Cannabis Use Problems?
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12/0278
Record Dates: First submitted 2014-01-22; First posted 2014-01-24 (Estimated); Last update posted 2018-10-24 (Actual); Status verified 2018-10

CONDITIONS: Cannabis Use Disorder
MeSH Terms: interventions — Cannabidiol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Cannabidiol 200mg Oral (Experimental)
  Interventions: Drug: Cannabidiol
- Cannabidiol 400mg Oral (Experimental)
  Interventions: Drug: Cannabidiol
- Cannabidiol 800mg Oral (Experimental)
  Interventions: Drug: Cannabidiol

INTERVENTIONS:
Drug: Cannabidiol
  Arms: Cannabidiol 200mg Oral; Cannabidiol 400mg Oral; Cannabidiol 800mg Oral
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this trial is to investigate a novel treatment for cannabis dependence: cannabidiol. Between 96 and 168 young people who want to quit cannabis and meet criteria for moderate cannabis use disorder (DSM-5) will be recruited from the community. Stage one aims to identify the Most Effective Dose (MEDmg) of oral cannabidiol for reducing cannabis use over four treatment weeks. Stage two will determine whether the MED identified in stage 1 can offer an effective treatment for cannabis dependence.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 16 and 60 years old.
* Meet DSM-5 criteria for moderate cannabis use disorder (≥4 DSM-5 criteria)
* Express desire to quit using cannabis within the next four weeks,
* Have ≥1 previous failed quit attempt.
* Smoke tobacco with cannabis,
* Test positive for recent cannabis use according to urine analysis,
* Vital signs within healthy limits and have capacity to give consent

Exclusion Criteria:

* Not willing to use effective contraception from when consent is taken to 6 weeks after treatment has stopped
* Positive pregnancy test or breastfeeding
* Allergies to the Investigational Medicinal Product (IMP) or placebo and its excipients
* >twice/month use of other illicit drugs
* Outside normal Body Mass Index (BMI)
* A physical health problem deemed clinically significant
* The use of current prescribed psychotropic drugs
* Current or prior self-reported diagnosis of a psychotic disorder
* Non-English speakers due to verbal assessments.

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 82 (Actual)
Dates: Start 2014-03; Primary Completion 2017-02-09 (Actual); Study Completion 2017-06-05 (Actual)

PRIMARY OUTCOMES:
Urinary 11-nor-9-Carboxy-delta-9-tetrahydrocannabinol:creatinine (THC-COOH:creatinine) | up to 4 weeks
  This study has two stages. This is the primary endpoint criteria for stage 1.
Number of days abstinent from cannabis | up to 4 weeks
  This study has two stages. This is the primary endpoint criteria for stage 1.
Diagnostic and Statistical Manual- 5 (DSM-5) criteria for moderate cannabis dependence | up to 4 weeks
  This study has two stages. This is the primary endpoint criteria for stage 2.
Urinary 11-nor-9-Carboxy-delta-9-tetrahydrocannabinol:creatinine(THC-COOH:creatinine) below 50ng/ml | week 4
  This study has two stages. This is the primary endpoint criteria for stage 2.

SECONDARY OUTCOMES:
Psychological Wellbeing, Cognition and Endocannabinoids | Up to 28 weeks
  Psychological Wellbeing, Cognition and Endocannabinoids will be measured by questionnaire methods, neuropsychological testing and biological samples.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Psychopharmacology Unit, London, United Kingdom

REFERENCES:
- [Derived] Lees R, Hines LA, Hindocha C, Baio G, Shaban NDC, Stothart G, Mofeez A, Morgan CJA, Curran HV, Freeman TP. Effect of four-week cannabidiol treatment on cognitive function: secondary outcomes from a randomised clinical trial for the treatment of cannabis use disorder. Psychopharmacology (Berl). 2023 Feb;240(2):337-346. doi: 10.1007/s00213-022-06303-5. Epub 2023 Jan 4. PMID 36598543
- [Derived] Freeman TP, Hindocha C, Baio G, Shaban NDC, Thomas EM, Astbury D, Freeman AM, Lees R, Craft S, Morrison PD, Bloomfield MAP, O'Ryan D, Kinghorn J, Morgan CJA, Mofeez A, Curran HV. Cannabidiol for the treatment of cannabis use disorder: a phase 2a, double-blind, placebo-controlled, randomised, adaptive Bayesian trial. Lancet Psychiatry. 2020 Oct;7(10):865-874. doi: 10.1016/S2215-0366(20)30290-X. Epub 2020 Jul 28. PMID 32735782